CLINICAL TRIAL: NCT03680664
Title: Enhancing Cognition in Older Persons: A Randomized Controlled Trial of Mindfulness-Based Stress Reduction (MBSR) and Transcranial Direct Current Stimulation (tDCS)
Brief Title: Mindfulness-Based Stress Reduction (MBSR) and Transcranial Direct Current Stimulation (tDCS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 065/2017
Record Dates: First submitted 2018-09-18; First posted 2018-09-21 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Anxiety Disorders; Mood Disorders; Transcranial Direct Current Stimulation; tDCS; Stress Reduction
Keywords: Mild Cognitive Impairment; Dementia; Mindfulness
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Cognitive Dysfunction; Dementia | interventions — Transcranial Direct Current Stimulation; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS + MBSR (Experimental): Excitatory bilateral stimulation to the frontal lobes, in particular the left and right DLPFC, will be applied. The anode will be placed at Fz and the cathode at Iz to achieve this bilateral frontal excitatory stimulation. Rubber electrodes will be inserted in 35-cm2 saline-soaked sponges and fixed with a headband. The direct current will be of 2 milliamps (mA) (current density = 0.57 A/m2) for 30 min per day.
  After a brief orientation session, the MBSR sessions will be conducted in 8 weekly 2.5 hour classes plus a half-day retreat. Content includes instruction and guidance to mindfulness meditation practices, gentle mindful movement, and various exercises to enhance mindfulness in everyday life. Participants will get daily at-home assignments with Compact Discs-Read Only Memory (CD-ROMs) of meditative practice.
  Interventions: Device: Active tDCS; Behavioral: MBSR
- sham tDCS + MBSR (Sham Comparator): The same tDCS parameters as as the active condition will be used; however, the device will be turned off after 1 minute of active stimulation.
  After a brief orientation session, the MBSR sessions will be conducted in 8 weekly 2.5 hour classes plus a half-day retreat. Content includes instruction and guidance to mindfulness meditation practices, gentle mindful movement, and various exercises to enhance mindfulness in everyday life. Participants will get daily at-home assignments with CDs of meditative practice.
  Interventions: Other: sham tDCS; Behavioral: MBSR

INTERVENTIONS:
Device: Active tDCS — Excitatory bilateral stimulation to the frontal lobes, in particular the left and right DLPFC, will be applied. The anode will be placed at Fz and the cathode at Iz to achieve this bilateral frontal excitatory stimulation. Rubber electrodes will be inserted in 35-cm2 saline-soaked sponges and fixed with a headband. The direct current will be of 2 mA (current density = 0.57 A/m2) for 30 min per day.
  Other Names: Transcranial Direct Current Stimulation
  Arms: Active tDCS + MBSR
Other: sham tDCS — The same tDCS parameters as as the active condition will be used; however, the device will be turned off after 1 minute of active stimulation.
  Arms: sham tDCS + MBSR
Behavioral: MBSR — After a brief orientation session, the MBSR sessions will be conducted in 8 weekly 2.5 hour classes plus a half-day retreat. Content includes instruction and guidance to mindfulness meditation practices, gentle mindful movement, and various exercises to enhance mindfulness in everyday life. Participants will get daily at-home assignments with CDs of meditative practice.
  Other Names: Mindfulness-Based Stress Reduction

SUMMARY:
Ideal interventions for the older aged population would be those that are easily accessible and associated with minimal burden on family members, the healthcare system and the individuals themselves. Mindfulness-Based Stress Reduction (MBSR) therapy and Transcranial Direct Current Stimulation (tDCS) are two interventions that may be effective in targeting cognitive deficits in individuals with anxiety, depression, and/or cognitive complaints. MBSR has been shown to decrease symptoms of depression and improve cognition and tDCS has been shown to improve cognition in the older aged population. The effectiveness of these two interventions combined to elicit changes in cognition has yet to be demonstrated. Therefore, the overall aim of the current research is to evaluate the efficacy of a combination of MBSR and tDCS to improve cognitive function in individuals with cognitive complaints and symptoms of anxiety and/or depression.

This will be a randomized pilot study. Sixteen individuals (separated into 2 groups of 8) will be randomized to receive a combination MBSR + active tDCS or MBSR + sham tDCS over 8 weeks. Participants will visit the Centre for Addiction and Mental Health (CAMH) once per week for in-class group sessions and will complete the intervention daily at home for the duration of the study. Participants will be aged 60 and older with cognitive complaints, with symptoms of anxiety and/or depression. Participants will be trained to self-administer tDCS and given guidelines for the completion of daily MBSR activities at home. It is hypothesized that the combination of active tDCS + MBSR will enhance cognition compared to the combination of sham tDCS + MBSR.

DETAILED DESCRIPTION:
Neurocognitive difficulties are a common problem in the older adult population. Previous research has shown memory complaints are higher in older adults with depression or anxiety versus those without these diagnoses. This suggests that mood symptoms, or a diagnosis of a mood disorder, may represent significant predictors of cognitive impairment. If left untreated, symptoms of depression and memory complaints may lead to greater cognitive impairment i.e. Mild Cognitive Impairment (MCI) and diagnosis of dementia . Therefore, early interventions are urgently needed to prevent decline in memory and cognitive function in individuals with MCI, depression, and/or anxiety.

This will be a randomized study design. Uo to 24 individuals (n=8 per group) will be randomized to receive a combination of 8-weeks of in-class group MBSR + active or sham tDCS and daily at-home MBSR + tDCS (active or sham). Each individual must be: (1) 60 or above; (2) present with cognitive complaints but not frank cognitive impairment (at a level of mild dementia or greater); and (3) present with a diagnosis or symptoms of depressed mood and/or anxiety.

Symptoms related to cognition, memory, and mood symptoms will be assessed at baseline (T0), throughout the study, as described in the MBSR protocol, and upon completion of the 8-week treatment course (Tx). Each study participant will have a clinical assessment at both T0 and Tx. Clinicians, participants and assessors will be blinded to the tDCS condition. These assessments will confirm any diagnoses and monitor clinical stability, including possible progression of participants to a diagnosis of a mood and/or anxiety disorder(s) or dementia. Any participant that progresses into a clinical diagnosis of dementia will be excluded from the study and referred to an appropriate level of care based on the severity of their symptoms.

To train participants on the tDCS intervention, each individual will attend one-week of in-class training sessions prior to initiating the 8-week study. Participants will come to the Centre for Addiction and Mental Health (CAMH) for 5 days leading up to the initiation of the MBSR treatment for tDCS self-administration training. On the final day of tDCS training, participants will attend a 2.5 hour in-class MBSR orientation session. Following this, the 8-week course of daily MBSR + tDCS will begin with an initial orientation session. The remaining 8 weeks of the at-home MBSR + tDCS intervention will be self-conducted at each participant's place of residence, with the exception of the weekly MBSR class each participant will be required to attend at CAMH. The study coordinator will be available by phone to the participants throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling men and women aged 60 or above.
2. Current cognitive complaints per participant self-report, but with intact cognitive function as defined by a score of 0-9 on the Short Blessed Test (SBT) and a Montreal Cognitive Assessment (MoCA) score ≥25 per PI discretion.
3. PROMIS depression scale score of greater or equal to 16 and/or PROMIS anxiety score greater or equal to 14.
4. Ability to read and speak English fluently enough to complete all research assessments.
5. Corrected visual ability to read newspaper headlines.
6. Hearing capacity to respond to a raised conversational voice.
7. Willingness and ability to provide informed consent.

Exclusion Criteria:

1. Diagnostic and Statistical Manual IV (DSM-IV) criteria for current or life-time bipolar disorder, schizophrenia, schizoaffective disorder or any other psychotic disorders.
2. Untreated post-traumatic stress disorder.
3. A MoCA score <25 or a score greater than 9 on the SBT, per PI discretion
4. Use of cognitive enhancers such as anticholinergic medications within the past 6weeks.
5. DSM-IV criteria for any substance dependence within the past 6 months that would affect their participation, per PI discretion.
6. Unstable medical illness (e.g. uncontrolled diabetes mellitus or hypertension).
7. Concurrent cognitive training, such as brain-training software, participation in psychotherapy or regular engagement in mindfulness practice and/or yoga.
8. Taking anticonvulsant or antipsychotics that cannot be safely tapered and discontinued.
9. Significant neurological condition (e.g. stroke, seizure disorder, multiple sclerosis).
10. A pace-maker or other metal implants that would preclude safe use of tDCS.
11. Intelligence Quotient (IQ) < 70 as estimated by the Wechsler Test of Adult Reading.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Change in cognitive and memory function | Baseline, Approximately 10-14 weeks after baseline
  Cognitive and memory function measured by a neuropsychological battery examining memory, executive functioning and attention

SECONDARY OUTCOMES:
Change in depressive symptoms | Baseline, Approximately 10-14 weeks after baseline
  Depressive symptoms as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) depressive symptoms
Change in anxiety symptoms | Baseline, Approximately 10-14 weeks after baseline
  Anxiety symptoms as as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) anxiety symptoms
Change in quality of life | Baseline, Approximately 10-14 weeks after baseline
  Quality of Life as assessed by PROMIS Scale for Ability to Participate in Social Roles and Activities, the PROMIS Scale for Satisfaction with Social Roles and Activities and the
Change in mindfulness | Baseline, Approximately 10-14 weeks after baseline
  Mindfulness as assessed by Cognitive Affective Mindfulness Scale - Revised (CAMS-R)

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Rajji, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Brooks H, Oughli HA, Kamel L, Subramanian S, Morgan G, Blumberger DM, Kloeckner J, Kumar S, Mulsant BH, Lenze EJ, Rajji TK. Enhancing Cognition in Older Persons with Depression or Anxiety with a Combination of Mindfulness-Based Stress Reduction (MBSR) and Transcranial Direct Current Stimulation (tDCS): Results of a Pilot Randomized Clinical Trial. Mindfulness (N Y). 2021;12(12):3047-3059. doi: 10.1007/s12671-021-01764-9. Epub 2021 Oct 5. PMID 34630733